CLINICAL TRIAL: NCT07357415
Title: A Phase 3b Study to Investigate the Efficacy and Safety of Different Retatrutide Dose Escalation Schemes in Participants Without Type 2 Diabetes Who Have Obesity or Overweight: A Randomized, Controlled, Double-Blind Trial
Brief Title: A Study of Retatrutide (LY3437943) in Participants Without Type 2 Diabetes Who Have Obesity or Overweight
Acronym: TRIUMPH-9
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27795; J1I-MC-GZQL (Other: Eli Lilly and Company)
Record Dates: First submitted 2026-01-16; First posted 2026-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — retatrutide

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Retatrutide Dose Escalation 1 (Experimental): Participants will receive retatrutide subcutaneously (SC)
  Interventions: Drug: Retatrutide
- Retatrutide Dose Escalation 2 (Experimental): Participants will receive retatrutide SC
  Interventions: Drug: Retatrutide
- Retatrutide Dose Escalation 3 (Experimental): Participants will receive retatrutide SC
  Interventions: Drug: Retatrutide

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of different retatrutide dose escalation schemes in participants without type 2 diabetes who have obesity or overweight. Participation in the study will last about 113 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a Body Mass Index (BMI) at screening

  * ≥ 30 kilogram per square meter (kg/m2) OR
  * ≥ 27 kg/m2 with presence of at least one of the following weight-related conditions at screening: high blood pressure, abnormal levels of lipid, obstructive sleep apnea, heart disease
* Have at least one unsuccessful attempt to lose weight by dieting

Exclusion Criteria:

* Have a self-reported change in body weight >5 kilograms (kg) (11 pounds) within 90 days before screening
* Have a prior or planned surgical treatment for obesity
* Have type 1 diabetes or type 2 diabetes
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have had within the past 90 days before screening:

  * heart attack
  * stroke
  * hospitalization for unstable angina or heart failure
* Have New York Heart Association Functional Classification Class IV congestive heart failure
* Have a history of chronic or acute pancreatitis
* Have taken weight loss drugs, including over-the counter medications within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-24 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 104

SECONDARY OUTCOMES:
Change from Baseline in Waist Circumference | Baseline, Week 104
Percent Change from Baseline in Triglycerides | Baseline, Week 104
Change from Baseline in Systolic Blood Pressure | Baseline, Week 104
Percent Change from Baseline in High Sensitivity C-Reactive Protein | Baseline, Week 104
Change from Baseline in Impact of Weight on Quality of Life-Lite-Clinical Trials (IWQOL-Lite-CT) Total Score | Baseline, Week 104
Overall Treatment Satisfaction with Medication for Obesity (TS-MO) Scores | Week 104
Pharmacokinetics (PK): Steady state Average Trough PK Concentration | Baseline through Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (20):
  - Arizona Research Center, Phoenix, Arizona
  - Care Access - Huntington Beach, Huntington Beach, California
  - Los Angeles Institute for Metabolic Research, Los Angeles, California
  - New Horizon Research Center, Miami, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - L-MARC Research Center, Louisville, Kentucky
  - Brigham and Women's Hospital Diabetes Program, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - NYC Research INC, Long Island City, New York
  - Weill Cornell Medical College, New York, New York
  - Care Access - Raleigh, Raleigh, North Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Cedar Health Research - Texas Native Health, Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - Cedar Health Research - Fort Worth, Fort Worth, Texas
  - Advanced Research Institute, Ogden, Utah
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - CAMC Institute for Academic Medicine, Charleston, West Virginia
- Argentina (5):
  - Cicemo Srl, Buenos Aires
  - CARDIAMET Investigaciones Médicas, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
- Canada (10):
  - Aggarwal and Associates Limited, Brampton
  - Med Trust Research, Courtice
  - Winterberry Research Inc., Hamilton
  - Diex Recherche Inc. Division Joliette, Joliette
  - Milestone Research Inc., London
  - Diex Recherche Inc. Division Quebec, Québec
  - Diex Recherche Inc. Division Sherbrooke, Sherbrooke
  - Canadian Phase Onward, Toronto
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto
  - C.I.C. Mauricie inc., Trois-Rivières

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in Participants Without Type 2 Diabetes Who Have Obesity or Overweight (TRIUMPH-9) — https://trials.lilly.com/en-US/trial/687735